CLINICAL TRIAL: NCT01423513
Title: Effects of Ankle Support on Muscle Activation and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: American Physical Therapy Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-16018
Record Dates: First submitted 2011-08-22; First posted 2011-08-26 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2012-04

CONDITIONS: Ankle Sprain
Keywords: ankle tape; Hoffmann reflex; Balance
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fibular Taping (Experimental): With the ankle in a neutral position, two strips of nonrigid hypoallergenic tape will be applied beginning at the distal aspect of the fibula, wrapping around the posterior aspect of the leg, and finishing superior and medial to the starting point. Next,a strip of rigid zinc oxide tape will be applied to the distal aspect of the fibula with tension.
  Interventions: Other: Fibular Taping
- Sham Taping (Sham Comparator): Sham taping will be applied in the same manner as the fibular taping, but tension will not applied to the zinc oxide tape
  Interventions: Other: Sham Taping

INTERVENTIONS:
Other: Fibular Taping — Tape with be applied with tension.
  Arms: Fibular Taping
Other: Sham Taping — Tape will be applied without tension
  Arms: Sham Taping

SUMMARY:
The purpose of this study is to examine the effects of ankle taping on improving muscle function and ankle motion in individuals who frequently twist (sprain) their ankle. It is thought that ankle taping may increase muscle function and ankle motion which would benefit individuals who frequently sprain their ankle.

DETAILED DESCRIPTION:
Previous research has demonstrated improved dynamic balance following the application of fibular taping. The effects of fibular taping on ankle dorsiflexion ROM and muscle activation in individuals with CAI are unknown. The purpose of this study is to determine the acute effects of fibular taping on muscle activation of the fibularis longus (peroneus) and soleus muscles, ankle dorsiflexion range of motion (ROM) and dynamic balance. The investigators hypothesize that fibular taping will have similar effectiveness as mobilization interventions which have been shown to improve muscle activation, ankle dorsiflexion ROM,and dynamic balance. Outcomes will be measured immediately before and after intervention. A crossover design will be used and participants will complete two visits at least 48 hours apart, but not more than 1 week apart. After participants complete both arms of the study their participation will be complete (average time to completion for each subject is 1 week).

ELIGIBILITY:
Inclusion Criteria:

* Age 16-45 years
* History of one or more ankle sprains
* Scoring at least an 85% on the Foot and Ankle Ability Measure (FAAM) Sport or at least 3 on the Modified Ankle Instability Instrument (AII).
* At least 5° ankle dorsiflexion asymmetry compared to the contralateral limb OR ankle dorsiflexion ROM less than 21°

Exclusion Criteria:

* Lower extremity injury or surgery within the past 6 months (including lateral ankle sprain)
* Diagnosed ankle osteoarthritis
* History of ankle surgery that involves intra-articular fixation
* Potential for current pregnancy

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Changes in muscle activation | All study visits up to day 7
  To determine the changes in muscle activation of the fibularis longus and soleus muscles following a fibular taping or sham taping intervention in individuals with CAI. Changes in muscle activation will be quantified by assessing the H-reflex technique before and after intervention.
  Hypothesis: We hypothesize that the fibular taping intervention will result in a greater activation of the fibularis longus and soleus muscles than a sham taping intervention.
Changes in ankle dorsiflexion range of motion (ROM) | All study visits up to day 7
  To determine the changes in ankle dorsiflexion ROM following a fibular taping or sham taping intervention in individuals with CAI. Changes in ankle dorsiflexion ROM will be quantified using a weight bearing lunge.
  Hypothesis: We hypothesize that the fibular taping intervention will result in a greater improvement in ankle dorsiflexion ROM than the sham taping intervention.
Changes in dynamic balance | All study visits up to day 7
  To determine the acute changes in balance following a fibular taping or sham taping intervention in individuals with CAI. Changes in balance will be quantified using the the Star Excursion Balance Test (SEBT).
  Hypothesis: We hypothesize that the fibular taping intervention will result in greater improvements in reach distance in all three SEBT directions compared to the sham taping intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton University, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Grindstaff TL, Hanish MJ, Wheeler TJ, Basnett CR, Miriovsky DJ, Danielson EL, Barr JB, Joseph Threlkeld A. Fibular taping does not alter lower extremity spinal reflex excitability in individuals with chronic ankle instability. J Electromyogr Kinesiol. 2015 Apr;25(2):253-9. doi: 10.1016/j.jelekin.2015.01.009. Epub 2015 Feb 16. PMID 25727519